CLINICAL TRIAL: NCT06903494
Title: Assessment of the 1-year Relapse Rate in Patients with Pemphigus Treated According to the Revised Pemphigus PNDS (national Diagnosis and Care Protocol)
Brief Title: Assessment of the 1-year Relapse Rate in Patients with Pemphigus Treated According to the Revised Pemphigus PNDS
Acronym: Etude PRERI
Status: Completed | Type: Observational
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Other Study IDs: 2020/144/OB; 2020-A01312-37 (Other: ANSM)
Record Dates: First submitted 2025-03-24; First posted 2025-03-30 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2024-03

CONDITIONS: Dermatology Disease
Keywords: pemphigus
MeSH Terms: conditions — Pemphigus

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
In May 2018, the PNDS (national diagnosis and care protocol) for pemphigus drawn up by the autoimmune bullous diseases reference centre was amended to take into account the results of recent studies and proposed, in line with the rituximab as 1st-line treatment: 1g repeated at 15-day intervals, then in the event of complete clinical remission, at 6 months: an infusion of 500mg or 1g in patients with initially severe pemphigus and/or who still have a high level of anti desmogleins at 3 months. The primary objective of the study is to prospectively evaluate the relapse rate during the first year of patients with newly diagnosed pemphigus treated according to the recommendations of the revised PNDS.

DETAILED DESCRIPTION:
Pemphigus is a rare, potentially life-threatening autoimmune bullous disease affecting both the skin and mucous membranes in which pathogenic IgG antibodies are directed against desmosomal transmembrane desmoglein (Dsg) 1 and 3. The initial severity of lesions in pemphigus correlates with levels of serum anti-Dsg antibodies anti-Dsg 1 and anti-Dsg 3 serum antibody levels, respectively. High doses of oral corticosteroids (OCs), sometimes combined with immunosuppressive drugs (azathioprine, mycophenolate mofetil) have been the mainstay of pemphigus treatment for many years for many years.

Over the last decade, more than 1,000 patients with recalcitrant or relapsing pemphigus have been treated pemphigus treated with rituximab (anti-CD20 monoclonal antibody) have been monoclonal antibody) have been reported in the literature.

The efficacy and safety of rituximab as a first-line treatment for patients with moderate to severe forms of pemphigus were recently evaluated in a large randomised controlled trial. Two predictive factors for early relapse that can be easily used in practice were identified, with a positive predictive value of 50% and a negative predictive value of 94% (initial PDAI severity score >45 and anti-desmoglein 1 >20 IU/ml and/or anti-desmoglein 3 >130 IU/ml at M3 after the first rituximab infusion).

Thus, the probability of an early relapse in patients presenting at least one of these 2 clinico-immunological criteria is 50%, whereas the probability of not relapsing in patients with none of these criteria is 94%.

In May 2018, the PNDS (national diagnosis and care protocol) for pemphigus drawn up by the autoimmune bullous diseases reference centre was amended to take into account the results of recent studies and proposed, in line with the rituximab as 1st-line treatment: 1g repeated at 15-day intervals, then in the event of complete clinical remission, at 6 months: an infusion of 500mg or 1g in patients with initially severe pemphigus and/or who still have a high level of anti desmogleins at 3 months. The primary objective of the study is to prospectively evaluate the relapse rate during the first year of patients with newly diagnosed pemphigus treated according to the recommendations of the revised PNDS.

ELIGIBILITY:
Inclusion Criteria:

1. Pemphigus newly diagnosed according to the following criteria:

   * erosions and/or superficial cutaneous and/or mucosal bullae, suggestive of pemphigus vulgaris (PV) or pemphigus superficialis (PS)
   * histological appearance of intraepidermal acantholysis
   * IgG and/or C3 deposits on the keratinocyte membrane (after meshwork)
2. Patient who has been informed
3. Moderate to severe pemphigus (PDAI score > 15), or mild pemphigus (PDAI score ≤ 15) that has not responded to the 1st line of treatment recommended in the NDSP (local corticosteroid therapy ± disulone) after three months.
4. Patient who has agreed to be monitored and treated according to the revised PNDS

Exclusion Criteria:

1. Patient âgé de moins de 18 ans
2. Diagnostic de Pemphigus (PV) ou (PS) restant incertain
3. Pemphigus paranéoplasique
4. Malade opposé à sa participation ou ne pouvant être suivi régulièrement

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients with newly diagnosed pemphigus treated as 1st-line patients with rituximab according to the recommendations of the revised PNDS,
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2021-02-17 (Actual); Primary Completion 2024-02-17 (Actual); Study Completion 2025-03-01 (Actual)

PRIMARY OUTCOMES:
Relapse rate over one year | 1 year
  The primary objective of the study was to prospectively evaluate the relapse rate during the first year of patients with newly diagnosed pemphigus treated according to the recommendations of the revised PNDS. Relapse' is defined as 'the reappearance of at least three new lesions per month, which do not heal spontaneously within one week or by the extension of old lesions in a patient who had previously achieved disease control.

SECONDARY OUTCOMES:
Evaluation of prognostic factors for short-term relapse (no maintenance infusion at 6 month)) | 6 month
  Determining no maintenance infusion at 6 month after after starting treatment by rituximab In patients with no risk factors for relapse .
Prognostic factors for short-term relapse (Tolerability of the treatment regimen proposed in the revised PNDS) | 1 year
  Assessment of severe and non-severe side effects during the 1st year of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Pascal PJ JOLY, Professor, Principal Investigator — University Hospital, Rouen
Locations (1):
- Pascal, Rouen, France

IPD SHARING:
Plan to Share IPD: No
The data provided will be the property of the sponsor and will be used solely for its own research activities.